CLINICAL TRIAL: NCT03938129
Title: Improving Women's and Children's Health Via Biobanking and Electronic Registry
Acronym: iELEVATE
Status: Completed | Type: Observational
Sponsor: Mark Santillan (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor-Investigator, Mark Santillan, Associate Professor, University of Iowa
Organization: University of Iowa (Other)
Other Study IDs: 201901749
Record Dates: First submitted 2019-05-02; First posted 2019-05-06 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Pregnancy Related; Maternal-Fetal Relations
MeSH Terms: interventions — Blood Specimen Collection; Pregnancy; Maternal Health

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 1st trimester maternal blood and urine sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: Pregnant women and their baby
  Interventions: Other: Blood sample; Other: Urine sample; Other: Pregnancy, maternal health, and fetal health data

INTERVENTIONS:
Other: Blood sample — 1st trimester blood sample for bio-bank
Other: Urine sample — 1st trimester urine sample for bio-bank
Other: Pregnancy, maternal health, and fetal health data — Pregnancy, maternal health, and fetal health data

SUMMARY:
Pregnancy related diseases and exposures in pregnancy are known risk factors for future disease. For example, women with a history of preeclampsia (a hypertensive disorder in pregnancy) and children born to these women are at increased risk of cardiovascular disease later in life. Yet, the mechanisms by which these long term health risks occur are unknown. Clearly, this presents a significant public health hazard as preventative and therapeutic interventions to block these pregnancy related diseases are limited. Current barriers to studying these long-term mechanisms in existing cohorts include 1) lack of paired long-term mother-child data, 2) lack of uniformly collected biosamples and 3) challenges in integrating data from multiple sources and institutions. In particular, data and biosample collection from rural and minority populations present significant challenges. The objective of the iELEVATE proposal is to expand and diversify a current biobank to accelerate long-term translational mechanistic and outcomes research in the vulnerable pregnancy population. We will accomplish this by establishing a widely available biorepository that will collect a first trimester blood and urine sample from pregnant women with a clinical data warehouse and e-registry to support long-term prospective cohort studies.

ELIGIBILITY:
Inclusion Criteria:

Pregnant women in their first trimester (less than 14 weeks) and have the capacity to provide informed consent are eligible to participate

Exclusion Criteria:

Under 18 years old, known non-viable pregnancy at time of consent,inability to provide informed consent and diagnosis of a known infectious disease.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pregnant woman in their first trimester.
Sampling Method: Non-Probability Sample
Enrollment: 1976 (Actual)
Dates: Start 2020-01-07 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
1.Number of Participants and Controls Enrolled in Biobank [ Time Frame: 2 years ] | 2 years
  Create bio-bank of maternal blood,urine and data.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Santillan, PhD, MD, Principal Investigator — University of Iowa
Locations (7):
- United States (7):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - OB Gyn Associates, PC, Cedar Rapids, Iowa
  - The Group Obstetrics & Gynecology Specialists, PC, Davenport, Iowa
  - University of Iowa, Iowa City, Iowa
  - West Des Moines OB GYN Associates, PC, West Des Moines, Iowa
  - University of Minnesota, Minneapolis, Minnesota
  - Marshfield Clinic Research Institute, Wausau, Wisconsin

IPD SHARING:
Plan to Share IPD: No